CLINICAL TRIAL: NCT04739111
Title: An Exploratory Clinical Study of Human Anti-PD-L1 Monoclonal Antibody Injection (LDP) Combined With Recombinant Anti-EGFR Human Mouse Chimeric Monoclonal Antibody Injection (CDP1) in Patients With Advanced Malignant Tumor
Brief Title: An Exploratory Clinical Study of LDP Combined With CDP1 in Patients With Advanced Malignant Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dragonboat Biopharmaceutical Company Limited (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCSW-LDP+CDP1-Ⅰ-01
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arms (Experimental): All participants will receive treatment with LDP combined with CDP1. In the dose-escalation phase, a fixed dose of CDP1 will be given once a week, while LDP will be given every two weeks with dose climbing. Then, cohort studies (cohorts 1 to 5) will be conducted during the dose-expansion phase.
  Interventions: Drug: Human Anti-PD-L1 Monoclonal Antibody Injection (LDP) Combined with Recombinant Anti-EGFR Human Mouse Chimeric Monoclonal Antibody Injection (CDP1)

INTERVENTIONS:
Drug: Human Anti-PD-L1 Monoclonal Antibody Injection (LDP) Combined with Recombinant Anti-EGFR Human Mouse Chimeric Monoclonal Antibody Injection (CDP1) — In the dose-escalation phase, CDP1 400 mg/ m2 will be given in the first week, then 250 mg/m2 will be given evert week. LDP will be given every two weeks with dose climbing of 5 mg/kg, 10 mg/kg, 20 mg/kg. Dose in the dose-expansion phase according to the assesment in the dose-escalation phase.
  Other Names: LDP combined with CDP1

SUMMARY:
This is an exploratory clinical study of Human Anti-PD-L1 Monoclonal Antibody Injection (LDP) combined with Recombinant Anti-EGFR Human Mouse Chimeric Monoclonal Antibody Injection (CDP1) in patients with advanced malignant tumor.

DETAILED DESCRIPTION:
This is an open, dose-escalation and dose-extension exploratory clinical study for patients with advanced malignancy who have failed standard therapy. In the dose-escalation phase, a fixed dose of CDP1 will be given once a week, while LDP will be given every two weeks with dose climbing. Then, cohort studies (cohorts 1 to 5) will be conducted during the dose-expansion phase. The purpose is to preliminarily evaluate the safety and efficacy of LDP combined with CDP1 in the treatment of patients with advanced malignant tumor, and to determine the recommended dose for clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 (inclusive), no gender limitation;
* 2. The estimated survival time is more than 3 months.
* 3. At least one assessable tumor lesion according to RECIST1.1 (in cohort 1, evaluate lesion is accept);
* 4. ECOG physical strength score 0-2;
* 5. No serious abnormal blood system, liver function, kidney function or coagulation function: ANC≥1.5×109 / L, PLT≥75×109 / L, Hb≥9g/dL; TBIL≤1.5×ULN, ALT≤2.5×ULN, AST≤2.5×ULN; Cr ≤ 1.5 × ULN, and creatinine clearance ≥ 50 ml /min(according to Croft Gault formula),Urinary protein ≤2+;or 24-hour urinary protein ≤1g; APTT≤ 1.5 ×ULN, PT ≤ 1.5 × ULN, INR ≤ 1.5 × ULN;"
* 6.Blood or urine pregnancy tests are negative in women of childbearing age within 7 days before the first dose.Male subjects and female subjects of reproductive age must use adequate contraception and have no plans to donate sperm or eggs within 3 months from the date of signing informed consent for the study to the date of the last study drug treatment.
* 7. Subjects must give informed consent to this study before the study, and voluntarily sign a written informed consent;
* 8.Locally advanced or metastatic malignancies diagnosed by histopathology, which have failed standard treatment, have no standard treatment regimen, or are not suitable for standard treatment at this stage. In the dose-expansion phase: cohort 1: head and neck squamous cell carcinoma;Cohort 2: colorectal cancer, RAS genotype was wild type;Cohort 3: esophageal squamous cell carcinoma;Cohort 4: Penile cancer;Cohort 5: Female reproductive system tumors (endometrial, cervical, ovarian).

Exclusion Criteria:

* 1. Received radiotherapy, chemotherapy, targeted therapy, endocrine therapy or immunotherapy within 4 weeks before the first administration, or other unlisted clinical trial drug therapy (mitomycin and nitrosourea are 6 weeks from the last administration, oral fluorouracil drugs such as tegiol and capecitabine are at least 2 weeks from the last administration, small molecule targeted drugs are at least 2 weeks or at least interval 5 half-life (Subject to the longer time) from the last administration, and traditional Chinese medicine with antitumor indications are at least 2 weeks from the last administration.
* 2. Major organ surgery (excluding puncture biopsy) or significant trauma occurred within 4 weeks prior to the first administration.
* 3. The adverse effects of previous antitumor therapy have not recovered to CTCAE 5.0 ≤grade1 (except for alopecia)
* 4. Patients with clinical symptoms of brain metastases, spinal cord compression, cancerous meningitis, or other evidence of uncontrolled brain or spinal cord metastases are not suitable for inclusion as judged by the investigator
* 5. Patients who had previously received PD-1 or PD-L1 inhibitors or anti-EGFR monoclonal antibody or other immune checkpoint inhibitors and failed;
* 6. Immunorelated adverse events ≥ Grade 3 were observed in previous immunotherapy;
* 7. Patients with active or previous autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, interstitial lung disease, etc.);
* 8. Patients who received systemic corticosteroid (prednisone > 10mg/ day or equivalent) or other immunosuppressive therapy within 14 days prior to initial dosing; Exceptions include: topical, ocular, intraarticular, intranasal, and inhaled corticosteroids;Short-term use of corticosteroids for preventive treatment;
* 9. Uncontrolled active hepatitis B (HBsAg positive with HBV DNA copy number > 103/ mL or HBV DNA titer >200 IU/ mL); Hepatitis C;Syphilis infection (syphilis antibody positive) and HIV positive patients.
* 10. A history of serious cardiovascular disease, including ventricular arrhythmias requiring clinical intervention;Acute coronary syndrome, congestive heart failure, stroke, or other grade 3 or higher cardiovascular events within 6 months;New York Heart Association (NYHA) cardiac function grade ≥II or left ventricular ejection fraction (LVEF) < 50%;Patients with clinically uncontrolled hypertension who are not suitable for the trial as determined by the investigator;
* 11. Known alcohol or drug dependence;
* 12. Mental disorder or poor compliance;
* 13. Women who are pregnant or lactating;
* 14. Have received live attenuated vaccine within 4 weeks before the first administration or scheduled to receive during the study period.
* 15. The Investigator considers that the subject is unsuitable to participate in this study because of any clinical or laboratory test abnormalities or other reasons.
* 16.A malignant tumor that has been active in the past two years (Except for tumors in this study, cured stage Ib cervical cancer or lower, non-invasive basal cell or squamous cell skin cancer, malignant melanoma with complete response (CR) > for 10 years, and other malignant tumors with complete response (CR) BBB>r 5 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From first dose of LDP combined of CDP1 through 30 days after last dose, up to 5 months.
  Adverse events (AEs) refer to all adverse medical events that occur when subjects sign the informed consent, which may be manifested as symptoms, signs, diseases or abnormal laboratory tests, but not necessarily causally related to the investigational drug.
Dose Limiting Toxicities (DLT) | Time Frame: 28 days after first dose of LDP combined of CDP1, up to 24 months.
  Number of participants with dose limiting toxicity (DLT)
Recommended dose for clinical trials | up to 24 months
  A comprehensive evaluation of the results from the dose escalation/expansion phase was conducted to determine the recommended dose for the clinical trial.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From first dose of LDP combined of CDP1, up to 2 years.
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Duration of response (DOR) | From first dose of LDP combined of CDP1, an average of 6 months.
  The duration of response (DOR) is defined as the time from the beginning of the first tumor assessment as PR or CR to the first assessment as PD or death from any cause.
Disease control rate (DCR) | From first dose of LDP combined of CDP1, up to 2 years.
  Disease control rate (DCR) is defined as the proportion of the optimal time response of CR, PR, disease stable (SD) (i.e. CR+PR+SD) between initiation of the trial drug and withdrawal from the trial, as assessed according to RECIST1.1 criteria
Progression-free survival (PFS) | From first dose of LDP combined of CDP1, an average of 6 months.
  Progression-free survival (PFS) is defined as the time elapsed from the day the study drug was first administered until the first imaging assessment of disease progression (PD) or death from any cause.
Maximum plasma concentrations (Cmax) | an average of 6 months
  Pharmacokinetic parameter, Observed Maximum Serum Concentration (Cmax) of LDP and CDP1.
Area under the plasma concentration-time curve from zero to last concentration time (AUC0-t) | an average of 6 months
  Pharmacokinetic Parameters, Area Under the Serum Concentration-time Curve From Time Zero to the Last Sampling Time (AUC0-t) of LDP and CDP1.
Half-life (t1/2) | an average of 6 months
  Pharmacokinetic parameters,Apparent Terminal Half-life (t1/2) of LDP and CDP1.
anti-drug antibody (ADA) | an average of 6 months
  Anti-drug antibody (ADA) is tested for immunogenicity assessment , titer and neutralizing antibody analysis were performed when ADA was positive, and immunocomplex (CIC) and complement analysis were performed.

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, Study Chair — West China Hospital
Locations (1):
- Dragonboat Biopharmaceutical,Co.,Ltd, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No